CLINICAL TRIAL: NCT02844426
Title: Effect of a Synbiotic on Symptoms of Patients With Slow Transit Constipation: A Prospective Randomized Trial
Brief Title: Effect of a Synbiotic on Symptoms of Patients With STC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Jianfeng Gong, Professor, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BIFICOPEC-2015
Record Dates: First submitted 2016-07-20; First posted 2016-07-26 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Slow Transit Constipation
Keywords: synbiotic; soluble dietary fiber; slow transit constipation; microbiota
MeSH Terms: interventions — Pectins; maltodextrin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): patients allowed to take maltodextrin by the experienced doctor.
  Interventions: Drug: maltodextrin
- synbiotic (Experimental): patients are allowed to take synbiotic (BIFICOPEC) contained 0.63g bifid triple viable capsule (BIFICO) and 8g soluble dietary fiber (Pectin) .
  Interventions: Drug: bifid triple viable capsule and pectin

INTERVENTIONS:
Drug: bifid triple viable capsule and pectin
  Arms: synbiotic
Drug: maltodextrin
  Arms: Placebo

SUMMARY:
To evaluate the efficacy of synbiotic (BIFICOPEC) containing Enterococci, Bifidobacteria, Lactobacilli triple viable bacteria and pectin in patients with slow transit constipation.

DETAILED DESCRIPTION:
Chronic constipation has become a common, often chronic, functional gastrointestinal disease which influences the quality of life all over the world. A total of 100 patients diagnosed as slow transit constipation (STC) using Rome III criteria were randomized to receive either synbiotic or placebo twice daily for 12 weeks. The primary efficacy endpoint was the clinical remission and improvement rate at week 4 and 12. Stool frequency and consistency, colonic transit time (CTT), evacuation and abdominal symptoms, Patient Assessment of Constipation Symptoms (PAC-SYM scores), Gastrointestinal Quality-of-Life Index (GIQLI), Satisfaction scores and adverse events were also monitored.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18 years;
2. BMI: 18.5-25kg/m2;
3. chronic constipation was diagnosed according to RomeⅢ criteria;
4. colonic transit time (CTT) >48 hours;
5. mild-to-moderate constipation with wexner constipation scale between 16 and 25.

Exclusion Criteria:

1. megacolon, intestinal obstruction, inflammatory bowel disease, and cancer;
2. secondary constipation (i.e. drugs, endocrine disorders, neurological disorders, metabolic disorders, psychological disorders or abdominal surgery);
3. severe anterior rectocele or full thickness rectorectal intussusception according to defecography;
4. pregnant or lactating women;
5. infection with enteric pathogen;
6. usage of antibiotics or proton pump inhibitors (PPIs);
7. hepatic, renal, cardiovascular, respiratory or psychiatric disease;
8. other diseases or factors evaluated by the investigator which could influence intestinal transit or intestinal microbiota.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-09; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Clinical remission rate | 3 months
  Patients having an average of three or more spontaneous complete bowel movements (SCBMs) per week were defined as remission.
Clinical improvement rate | 3 months
  Patients with an average increase of one or more spontaneous complete bowel movements (SCBMs) per week were defined as improvement.

SECONDARY OUTCOMES:
Number of bowel movements per week | 3 months
Stool consistency according to the Bristol Stool Form Scale (BSFS) | 3 months
  Stool types 1 and 2 indicated constipation; types 3, 4, and 5 indicated normal; and types 6 and 7 indicated diarrhea.
Colonic transit time (CTT) | 3 months
  CTT was measured by Metcalf method.
Patient Assessment of Constipation Symptoms (PAC-SYM) questionnaire | 3 months
  The questionnaire contained 12 symptoms which were grouped into three subscales for stool, abdominal and rectal symptoms.
The Gastrointestinal Quality-of-Life Index (GIQLI) | 3 months
  To evaluate specific quality of life in patients with gastrointestinal diseases, comprised 36 questions using a 5-point Likert-type scale ranging from 0 to 4 (0, worst; 4, best).
Satisfaction score of constipated patients | 3 months
  The score ranged from 1 (extremely unsatisfied) to 5 (extremely satisfied).
Abdominal symptoms | 3 months
  Patients recorded their symptoms of abdominal pain or cramps and bloating or flatulence according to five classifications of symptoms (1, none; 2, mild; 3, moderate; 4, severe; 5, very severe).
Evacuation symptoms | 3 months
  Patients recorded their perception of straining, lumpy hard stools, sensation of incomplete evacuation, and sensation of anorectal blockage according to a 5-point ordinal scale (1, none; 2, mild; 3, moderate; 4, severe; 5, very severe).
Treatment-related adverse events | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, Study Director — department of generay surgery, jinling hospital
Locations (1):
- Department of Generay Surgery, Jinling hosptal, Medical School of Nanjing University, Nanjing, Jiangsu, China